CLINICAL TRIAL: NCT03356587
Title: A Biomarker-driven, Open Label, Single Arm, Multicentre Phase II Study of Abemaciclib in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Who Failed to Platinum-based Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13Y-MC-E011
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-09

CONDITIONS: HNSCC; Head and Neck Neoplasms
Keywords: NGS; Nanostring; Biomarker Driven Umbrella Trial; abemaciclib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: During or after palliative 1st line platinum based chemotherapy, we will perform prescreening NGS based molecular characterization.
  Molecular tumor board to determine characterization will be held for every patients. Once each patients have relevant genetic pathway, the patients will be allocated each treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm4: Abemaciclib (Experimental): Abemaciclib represents a selective and potent small molecule CDK4 and CDK6 dual inhibitor with broad antitumor activity in preclinical pharmacology models.(oral class) Patients will be instructed to take Abemaciclib orally at a dose of 200mg bid with a glass of water twice daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Patients will be instructed to take Abemaciclib orally at a dose of 200mg bid with a glass of water twice daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day

SUMMARY:
Open, multicenter, single arm, phase II, biomarker driven umbrella trial for head and neck squamous cell carcinoma (FGFR inhibitor, CDK4/6 inhibitor, pan HER inhibitor, PI3K inhibitor, PD1/PD-L1 inhibitor)

DETAILED DESCRIPTION:
This study will be conducted as a treatment arm 4 of the umbrella clinical trial.(NCT03292250)

During or after palliative 1st line platinum based chemotherapy, we will perform prescreening NGS based molecular characterization. The molecular characterization will be done by following three methods.

* NGS : Agilent SureSelect Target Enrichment (245 genes)
* Nanostring nCounter including immune signature
* IHC : PD-L1

The present trial will investigate the efficacy and safety of abemaciclib in patients with recurrent or metastatic HPV (-) HNSCC with genetic alterations of cell cycle pathway who failed to platinum-based therapy. We will also evaluate feasibility and the effect on decision making of next generation sequencing of HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* (1) Histologically or cytologically confirmed recurrent or metastatic HNSCC, except nasopharyngeal carcinoma (2) Age ≥20 (3) ECOG performance status of 0-1 (4) Ineligibility for local therapy (surgery or radiotherapy) (5) Prior palliative chemotherapy including platinum-based chemotherapy. When recurred within 6 months of definitive/neoadjuvant/adjuvant chemo- or chemoradiation, the chemotherapy is considered a line of palliative chemotherapy (6) At least one measurable lesion by RECIST ver 1.1 (7) p16 negative and intact Rb and genetic alterations in CDK4/6 pathway (8) Adequate organ function for all of the following criteria, as defined below.
* Absolute neutrophil count (ANC) ≥1500 cells/mm3
* Platelets ≥100,000 cells/mm3
* Hemoglobin ≥ 8 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
* Serum creatinine ≤1.5 x institution upper limit of normal
* Total Bilirubin ≤1.5 x upper limit of normal (ULN) (Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.)
* AST (SGOT) ≤3.0 x ULN
* ALT (SGPT) ≤3.0 x ULN (9) If a female of childbearing potential, must have a negative serum pregnancy test within 7 days of the first dose of abemaciclib and agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of abemaciclib.

If a male, must agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following the last dose of abemaciclib. Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.

(10) Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to screening. A washout period of at least 21 days is required between last chemotherapy dose and screening (provided the patient did not receive radiotherapy).

(11) Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.

(12) The patient has provided signed informed consent and has a compliance to follow the study protocol.

(13) The patient is able to swallow oral medications.

Exclusion Criteria:

* (1) Prior treatment with CDK4/6 pathway inhibitors (2) Nasopharyngeal carcinoma (3) The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).

  (4) Pregnant woman, Breast-feeding woman (5) Recent significant bleeding history within 6 major vessel invasion of tumor (6) Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial (infection/inflammation, intestinal obstruction, social/psychological complications).

  (7) Patient who have an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies) (8) The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | 24 months
  RECIST version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  RECIST version 1.1
Overall survival (OS) | 24 months
  Overall Survival is defined as the time from first dose to death due to any cause. Through the follow-up within 30 days after study completion or termination of the last subject, death and date of death will be checked for subject alive during treatment period
Duration of response | 24 months
  RECIST version 1.1
Toxicity | 24 months
  number of patients with treatment-related AE as assessed by NCI CTCAE version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
anticipated as research paper